CLINICAL TRIAL: NCT06686862
Title: Non-Steroidal Anti-Inflammatory Drugs Versus Conventional Treatment in Acute Myocarditis (INFLAMA Trial)
Brief Title: Non-Steroidal Anti-Inflammatory Drugs in Acute Myocarditis
Acronym: INFLAMA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Collaborators: Fundación Investigación Biomédica Puerta de Hierro Majadahonda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-513803-15-00; 2024-513803-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-02

CONDITIONS: Myocarditis Acute
Keywords: Nonsteroidal antiinflammatory agents; Magnetic Resonance Imaging
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The analysis of the cardiac magnetic resonance imaging will be performed by evaluators blinded to the treatment and the timing of the imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen (Experimental): Ibuprofen tapering schedule during 3 weeks.
  Interventions: Drug: ibuprofen
- Acetaminophen (No Intervention): Acetaminophen or metamizole in case of allergy until pain resolution, according to routine clinical practice.

INTERVENTIONS:
Drug: ibuprofen — Ibuprofen tapering schedule during 3 weeks. First week: Ibuprofen 600 mg every 8 hours. Second week: Ibuprofen 600 mg every 12 hours. Third week: Ibuprofen 600 mg every 24 hours.
  Arms: Ibuprofen

SUMMARY:
Prospective, randomized, multicenter, open-label clinical trial to evaluate the safety and efficacy of a 3-week ibuprofen tapering regimen compared to conventional analgesic treatment (acetaminophen) in patients with acute myocarditis and left ventricular ejection fraction ≥50%. The objective is to assess the reduction in late gadolinium enhancement on cardiac magnetic resonance imaging at 6-month follow-up.

DETAILED DESCRIPTION:
The treatment for patients with uncomplicated myocarditis (left ventricular ejection fraction >50% without heart failure) is not currently well defined. Analgesic drugs are commonly used to manage pain. The use of nonsteroidal anti-inflammatory drugs (NSAIDs) among analgesics is controversial due to potential harmful effects observed in animal models. However, NSAIDs are the standard treatment for pericarditis, even when it is associated with mild myocardial involvement. In patients with acute myocarditis and normal left ventricular ejection fraction, observational studies have suggested that NSAIDs may have a beneficial effect in reducing late gadolinium enhancement (LGE) measured in cardiac magnetic resonance (CMR), an important prognostic marker in this population.

We plan to conduct a prospective, randomized, multicenter, open-label clinical trial to evaluate the safety and efficacy of NSAIDs versus conventional analgesic treatment in patients with uncomplicated acute myocarditis and left ventricular ejection fraction ≥50%.

Approximately 150 patients will be randomized 1:1 to NSAID treatment (ibuprofen tapering schedule during 3 weeks) or conventional treatment (acetaminophen or metamizole in case of allergy until pain resolution) during hospital admission. Patients will be followed for a 12-month period. Baseline CMR will be performed at initial hospitalization for acute myocarditis and at 3 and 6 months.

The primary objective is to assess the utility of ibuprofen versus conventional treatment with analgesics in acute myocarditis with preserved LVEF, in terms of reducing LGE on CMR at 6-month follow-up compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Patients hospitalized for confirmed acute myocarditis and left ventricular ejection fraction ventricular >50%.
* Elevated troponin I/T (3 times above the upper limit of normal).
* Absence of acute heart failure.
* Absence of ischemic heart disease (ruled out by coronary angiography or coronary CT in individuals over 40 years).
* Diagnostic criteria for myocarditis (Lake Louise, 2018 update) by cardiac magnetic resonance imaging.

Exclusion Criteria:

* Kidney disease stage 3b, 4 and 5 (creatinine clearance by CKD-EPI <45 ml/min/1.73 m2).
* Severe liver failure (Child-Pugh class C).
* Poorly controlled pharmacological hypertension (repeatedly systolic arterial pressure >140 mmHg).
* Diagnosis criteria for acute pericarditis.
* Moderate or severe pericardial effusion (>10 mm in total).
* Hypersensitivity to NSAIDs or previous use in the last 7 days.
* Contraindication for MRI.
* Participation in another clinical trial.
* Pregnancy, breastfeeding, or women of childbearing age unwilling to use appropriate contraception throughout the study.
* Any circumstance that, in the investigator's opinion, compromises participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in late gadolinium enhancement (measured in % relative to indexed myocardial mass) compared to baseline (CMR) at admission) | 6 months

SECONDARY OUTCOMES:
Change in late gadolinium enhancement (measured in % relative to indexed myocardial mass by CMR) compared to baseline at 3 months. | 3 months
Changes in T2 mapping values (measured in milliseconds by CMR) compared to baseline at 6 months. | 6 months
Changes in T2 mapping values (measured in milliseconds by CMR) compared to baseline at 3 months. | 3 months
Changes in T1 mapping values (measured in milliseconds) and extracellular volume (measured in %) by CMR compared to baseline at 6 months. | 6 months
Changes in T1 mapping values (measured in milliseconds) and extracellular volume (measured in %) by CMR compared to baseline at 3 months. | 3 months
Compare exercise capacity using METs (metabolic equivalent) in conventional treadmill exercise test at 3 months. | 3 months
Proportion of patients experiencing arrhythmias during treadmill exercise test at 3 months | 3 months
Proportion of patients from each group experiencing hospitalization due to recurrent myocarditis, heart failure, severe ventricular arrhythmias, or cardiovascular death at 12 months. | 1 year
Proportion of patients developing adverse events in each treatment group at 1 month | 1 month
  Adverse events: severe adverse event, grade 3-4 adverse event, adverse reaction, special interest adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Domínguez-Rodriguez, MD, PhD, Principal Investigator — Heart Failure and Inherited Cardiac Diseases Unit, Department of Cardiology, Hospital Universitario Puerta de Hierro, IDIPHISA, Madrid, Spain; Pablo García-Pavía, MD, PhD, Principal Investigator — Heart Failure and Inherited Cardiac Diseases Unit, Department of Cardiology, Hospital Universitario Puerta de Hierro, IDIPHISA, Madrid, Spain
Locations (1):
- Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under agreement, individual or aggregated patient data could be shared with other scientific groups for scientific projects. Data can be shared only for scientific purposes and in full compliance with Personal Data Protection requirements in the EU.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study scientific publication
Access Criteria: Under request to Study Chair